CLINICAL TRIAL: NCT05593341
Title: Effect of Perioperative Opioid Education on Outcomes After Total Knee Arthroplasty: A Randomized Study
Brief Title: Opioid Education in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-1286
Record Dates: First submitted 2022-09-30; First posted 2022-10-25 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Arthropathy of Knee; Post Operative Pain; Opioid Use; Opioid Abuse; Opioid Misuse
Keywords: Opioid Education
MeSH Terms: conditions — Pain, Postoperative; Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Patients are referred to the Hospital's standard 1-hour virtual patient education webinar prior to surgery.
- In-person and PDF (Experimental): Patients will receive two in-person education sessions (1st session before surgery and 2nd session after surgery). Patients will also receive pdf handouts about opioids and pain management.
  Interventions: Other: Opioid education in person
- Video and PDF (Experimental): Patients will receive two video education sessions (1st session before surgery and 2nd session after surgery). Patients will also receive pdf handouts about opioids and pain management.
  Interventions: Other: Opioid education via video

INTERVENTIONS:
Other: Opioid education in person — The presentation and handouts contain information regarding the following topics:
  * Reviewing opioids and strategies for analgesia
    * Defining and identifying opioids
    * Goals for postoperative pain management and utilizing opioids to treat pain
    * Alternative modes of treating pain
    * Regional anesthesia/analgesia defined
  * Side effects and risks of opioids
    * Common side effects of opioids
    * Risks of addiction, tolerance, dependence, opioid-induced hyperalgesia with long-term use
  * Proper use and handling of opioids
    * Safe practices when taking opioids
    * Weaning off opioids
    * Safe storage and disposal of opioids
  Arms: In-person and PDF
Other: Opioid education via video — The video and handouts contain information regarding the following topics:
  * Reviewing opioids and strategies for analgesia
    * Defining and identifying opioids
    * Goals for postoperative pain management and utilizing opioids to treat pain
    * Alternative modes of treating pain
    * Regional anesthesia/analgesia defined
  * Side effects and risks of opioids
    * Common side effects of opioids
    * Risks of addiction, tolerance, dependence, opioid-induced hyperalgesia with long-term use
  * Proper use and handling of opioids
    * Safe practices when taking opioids
    * Weaning off opioids
    * Safe storage and disposal of opioids
  Arms: Video and PDF

SUMMARY:
The goal of this experimental study is to compare different education intervention on opioid education for patients undergoing total knee arthroplasty. The specific research questions to address are:

1. Does perioperative education pathway reduce opioid refill requests?
2. Is education pathway that focuses on pain management provided in-person and via video in repeated sessions more effective than current standard of care education consisting of a single exposure given as part of a broader preoperative presentation covering multiple topics?
3. Is there a difference between education provided in-person vs video?
4. Does perioperative education improve compliance with multimodal analgesia?
5. Does perioperative education improve appropriate opioid storage?
6. Does perioperative education improve appropriate opioid disposal?

Enrolled patients will be assigned at random to one of 3 study groups. Group 1 (control): Patients are referred to the hospital's standard 1-hour virtual patient education webinar prior to surgery.

Group 2 (in-person): Patients will receive two in-person education sessions (1st session before surgery and 2nd session after surgery). Patients will also receive portable document format (pdf) handouts about opioid and pain management.

Group 3 (video): Patients will receive two video education sessions (1st session before surgery and 2nd session after surgery). Patients will also receive pdf handouts about opioid and pain management.

DETAILED DESCRIPTION:
Patients undergoing surgery are frequently unaware of how to properly use opioids for pain management which may result in poor compliance with pain regimens, worse pain control and functional outcomes, and improper storage and disposal. There is evidence that educational interventions in various formats may improve pain and promote proper opioid handling. In addition, multimodal analgesia has been shown to be effective in total joint arthroplasty, and setting appropriate expectations may reduce anxiety, postoperative recovery time, and post surgical acute pain.

The current education process at HSS involves patient referral to a virtual webinar which is optional. Pain topics are covered within a broader 50-minute presentation on numerous topics related to surgery. Information on pain topics may be difficult to process and retain because it is a single exposure that is combined with multiple unrelated topics, and there is no repetition or reference provided. The aim of this study is to explore how a comprehensive educational pathway focusing on aspects of pain control and proper opioid use with repeated sessions will affect outcomes after total knee arthroplasty by comparing three groups - 1) patients who attend the virtual webinar, 2) an in-person session with a portable document format (PDF), and 3) a video session with PDF.

ELIGIBILITY:
Inclusion Criteria:

* Age between age 18 and 80 years old
* Undergoing primary total knee replacement surgery at Hospital for Special Surgery
* English speaking

Exclusion Criteria:

* History of chronic opioid use (continuous opioid use for 3 or more months)
* Opioid use within the past 3 months
* Contraindication to NSAIDs or acetaminophen
* Contraindication or allergy to opioids
* Contraindication to any study medications (i.e., fentanyl, ketamine, versed, acetaminophen, ketorolac, zofran, decadron)
* Discharge to rehab or skilled nursing facility (opioids are not prescribed by HSS providers)
* Contraindication or refusal to receive neuraxial anesthesia or peripheralnerve blocks (PNB)
* Revision surgery
* Ambulatory surgery
* Patients who are pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Opioid refill at POD 30 | Post operative day (POD) 30
  Patients will be asked if they have refilled their opioid prescription and the number of opioid refills.
Opioid refill at POD 60 | Post operative day (POD) 60
  Patients will be asked if they have refilled their opioid prescription and the number of opioid refills.

SECONDARY OUTCOMES:
Hospital length of stay | From the time patient enters the post-anesthesia care unit (PACU entry) until the time patient is discharged from the hospital (discharge time), assessed up to 168 hours (1 week)
  The total amount of time spent in-patient following their surgery.
Patient's health and recovery status following their surgery | Pre-operative (when patient is in the holding area being prepped for surgery), Post-operative day 1, Post-operative day 7, Post-operative day 14
  A survey titled: quality of recovery 15 (QoR15) is a patient- reported outcome measure measuring quality of recovery after surgery and anesthesia.
  Each of the following question on the survey will be assessed on a 0-10 scale, with 0 meaning "none of the time" and 10 meaning "all of the time".
  How have you been feeling in the last 24 hours?
  1. Able to breathe easily
  2. Been able to enjoy food
  3. Feeling rested
  4. Have had a good sleep
  5. Able to look after personal toilet and hygiene unaided
  6. Able to communicate with family or friends
  7. Getting support from hospital doctors and nurses
  8. Able to return to work or usual home activities
  9. Feeling comfortable and in control
  10. Having a feeling of general well-being
      Have you had any of the following in the last 24 hours?
  11. Moderate pain
  12. Severe pain
  13. Nausea or vomiting
  14. Feeling worried or anxious
  15. Feeling sad or depressed
Numerical Rating Scale | Post-operative day 0, Post-operative day 1, Post-operative day 7, Post-operative day 14
  Patients are asked to report a number between 0 and 10 that best measures their pain intensity. Zero represents 'no pain at all' whereas 10 represents 'the worst pain ever possible'.
Opioid consumption | Post-operative day 0, Post-operative day 1, Post-operative day 7, Post-operative day 14
  The amount of opioid consumption by the patient (in oral morphine equivalents).
Rates of compliance with multimodal regimen | Post-operative day 1, Post-operative day 7, Post-operative day 14
  Patients will keep "pain diary" to record use of each medication (acetaminophen, NSAIDs, and opioid). Compliance will be defined as the percentage of prescribed medication (acetaminophen or NSAID) that is actually taken.
Rates of proper opioid storage | Post-operative day 7
  Patients will be asked to report how they are storing their opioids (i.e., stored "locked and hidden").
Rates of proper opioid disposal | Post-operative day 21
  Patients will be asked to report how they are disposing of their unused opioids (i.e., reporting they dispose using one of the accepted proper disposal methods).

CONTACTS AND LOCATIONS:
Overall Officials: Bradley H Lee, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.

REFERENCES:
- [Result] Lee BH, Wu CL. Educating Patients Regarding Pain Management and Safe Opioid Use After Surgery: A Narrative Review. Anesth Analg. 2020 Mar;130(3):574-581. doi: 10.1213/ANE.0000000000004436. PMID 31567320
- [Result] Syed UAM, Aleem AW, Wowkanech C, Weekes D, Freedman M, Tjoumakaris F, Abboud JA, Austin LS. Neer Award 2018: the effect of preoperative education on opioid consumption in patients undergoing arthroscopic rotator cuff repair: a prospective, randomized clinical trial. J Shoulder Elbow Surg. 2018 Jun;27(6):962-967. doi: 10.1016/j.jse.2018.02.039. Epub 2018 Mar 26. PMID 29599038
- [Result] Egan KG, De Souza M, Muenks E, Nazir N, Korentager R. Opioid Consumption Following Breast Surgery Decreases with a Brief Educational Intervention: A Randomized, Controlled Trial. Ann Surg Oncol. 2020 Sep;27(9):3156-3162. doi: 10.1245/s10434-020-08432-7. Epub 2020 Apr 13. PMID 32285282
- [Result] Horn A, Kaneshiro K, Tsui BCH. Preemptive and Preventive Pain Psychoeducation and Its Potential Application as a Multimodal Perioperative Pain Control Option: A Systematic Review. Anesth Analg. 2020 Mar;130(3):559-573. doi: 10.1213/ANE.0000000000004319. PMID 31335400
- [Result] Memtsoudis SG, Poeran J, Zubizarreta N, Cozowicz C, Morwald EE, Mariano ER, Mazumdar M. Association of Multimodal Pain Management Strategies with Perioperative Outcomes and Resource Utilization: A Population-based Study. Anesthesiology. 2018 May;128(5):891-902. doi: 10.1097/ALN.0000000000002132. PMID 29498951
- [Result] Stepan JG, Sacks HA, Verret CI, Wessel LE, Kumar K, Fufa DT. Standardized Perioperative Patient Education Decreases Opioid Use after Hand Surgery: A Randomized Controlled Trial. Plast Reconstr Surg. 2021 Feb 1;147(2):409-418. doi: 10.1097/PRS.0000000000007574. PMID 33235041
- [Result] Nahhas CR, Hannon CP, Yang J, Gerlinger TL, Nam D, Della Valle CJ. Education Increases Disposal of Unused Opioids After Total Joint Arthroplasty: A Cluster-Randomized Controlled Trial. J Bone Joint Surg Am. 2020 Jun 3;102(11):953-960. doi: 10.2106/JBJS.19.01166. PMID 32251139
- [Result] Osterberg L, Blaschke T. Adherence to medication. N Engl J Med. 2005 Aug 4;353(5):487-97. doi: 10.1056/NEJMra050100. No abstract available. PMID 16079372
- [Derived] Sheetz M, Puglisi A, Trentalange M, Reichel J, Chalmers B, Gonzalez Della Valle A, Sideris A, Lee BH. Comparing modalities of opioid education in patients undergoing total knee arthroplasty: a randomized pilot trial. Reg Anesth Pain Med. 2026 Jan 5;51(1):60-68. doi: 10.1136/rapm-2024-105701. PMID 39327049

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT05593341/Prot_SAP_000.pdf